CLINICAL TRIAL: NCT04062838
Title: Prospective Pilot Study: Prolotherapy For The Treatment Of Patients With Partial Rotator Cuff Tears
Brief Title: Prolotherapy for the Treatment of Partial Rotator Cuff Tears
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: I did not receive funding to finance this study
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0391-18-HMO
Record Dates: First submitted 2018-08-01; First posted 2019-08-20 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2020-05

CONDITIONS: Rotator Cuff Tear
Keywords: partial; prolotherapy; subacromial steroid injection; tendon healing; tendon tear enlargement
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Glucose; Solutions

STUDY DESIGN:
Intervention Model Description: The aim of this trial is to study the effects of injected glucose on injured or degenerative rotator cuff tears of the shoulder. Glucose is not recognised by the FDA for this purpose but is used in 2 main concentrations: 50% solution to treat hypoglycemia and 5% solution for fluid replacement.
Masking Description: evaluating radiologist will all be blinded to the dates of the scans.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prolotherapy (Experimental): Injection of 20% dextrose (50 % dextrose diluted with 0.5% lidocaine) into the rotator cuff tendinous insertions as well as into the tear. All injections are performed under ultrasound.
  Interventions: Drug: Dextrose 50

INTERVENTIONS:
Drug: Dextrose 50 — As above
  Other Names: Glucose 50% solution

SUMMARY:
This is a Prospective Pilot Single Arm study on prolotherapy for the treatment of patients with pain due to Partial Rotator Cuff (RC) Tears of the Shoulder.

The aim of this trial is to study the effects of injected glucose on injured or degenerative RC tears of the shoulder. Glucose is not recognized by the FDA for this purpose but is used in 2 main concentrations: 50% solution to treat hypoglycemia and 5% solution for fluid replacement.

In the prolotherapy group, 20% dextrose will be injected into 4 locations of the affected shoulder. In the active control group, patients will receive a single injection of methylprednisolone into the subacromial bursa and 3 saline injections overlying the tendons.

DETAILED DESCRIPTION:
Prolotherapy treatments have been used since the 1950s for the treatment of weakened or damaged soft tissue and cartilage. Pre-clinical studies have demonstrated an anabolic response leading to thickened collagen tissue following treatment. Prolotherapy has been used to treat various tendinopathies, non-specific low back pain whiplash injuries, and partial ligament and tendon tears. Injection solutions used in the past include P2G (phenol, glycerine and glucose), sodium morrhuate and simple dextrose. Today, most prolotherapists use simple dextrose as an off-label treatment. Current treatment methods of the RC have several short-comings. Steroid injections, the most commonly applied treatment today for RC tears, have a short term benefit at the very most and have been found, when repeated, to lead to deterioration in pain, function and even tendon structure. Surgery is expensive, requires a long rehabilitation program, and has a very significant re-tear rate. In addition, studies are not conclusive regarding its effectiveness as compared to conservative treatment for the treatment of RC tears. No prolotherapy studies have been performed in the treatment of partial RC tears. Considering the extent of this endemic disorder, it was decided to explore prolotherapy for the treatment of partial rotator cuff tears.

• Patients will be referred from local community clinics both by orthopedic surgeons as well as from family physicians. Patients will have received a steroid injection into the subacromial bursa and will have failed to respond.

Patients will receive 3 monthly treatments all under ultrasound.

25 patients will be recruited to this Pilot study. It is impossible to make an accurate estimation of the sample size of the trial needed as no prolotherapy study has been done specifically on partial RC tears.

* Patients with partial tears of less than 1 cm measured in a thorough ultrasound examination either in length or in width in any of the rotator cuff tendons are eligible for the trial.
* Patients will sign a consent form. They will rate their pain NRS score out of 10 prior to treatment and fill out (hopefully) an Oxford Shoulder Score (OSS) Questionnaire. (The principle investigator has translated this questionnaire into Hebrew and has received approval from Oxford University for use in this research).
* Dr. Wende will perform all treatments under ultrasound in both groups, up to 3 treatments in each patient.
* The radiologist evaluating pre and post treatment ultrasound scans will be blinded to the dates of the exam.
* Before the first treatment, an ultrasound scan of the shoulder will be performed by a musculoskeletal radiologist in Hadassah.
* 4 points within the shoulder will be injected. Structures to be injected will include the supraspinatus, infraspinatus and subscapularis tendons as well as the inferior glenohumeral ligament. 20% dextrose and 0.5% lidocaine will be injected.
* All patients will be followed up by an unbiased, independent investigator 1, 6 and 12 months after the last treatment at which time the NRS pain score is questioned and an OSS questionnaire is filled out.
* 6 months after the last treatment, patients will have a repeat ultrasound scan of the shoulder 6 and 12 months after the last treatment, the range of shoulder motion will be examined by an independent investigator.

ELIGIBILITY:
Inclusion Criteria:

* With partial rotator cuff tears of either the supraspinatus, infraspinatus or subscapularis tendons of less than 1cm in either length or width
* With pain lasting more than 6 months
* Pain with an NRS score of at least 6 out of 10

Exclusion Criteria:

* Who had surgical repair, arthroscopy of the affected shoulder
* With rotator cuff tears larger than 1cm
* With Rotator cuff arthropathy or osteoarthritis of the glenohumeral joint
* With primary adhesive capsulitis (frozen shoulder secondary to partial RC tear is not an exclusion criterion)
* With active malignant disease
* With fibromyalgia or depression, the latter significant enough to affect their daily life
* With a history of inflammatory joint disease
* With localized (to the involved arm) or generalised neuropathic pain
* With a history of bone fracture within the shoulder girdle which is still causing pain
* Currently medicated with corticosteroids
* With active infection
* Who smoke either tobacco or cannabis
* Who are pregnant
* With uncontrolled diabetes
* Who have any contra-indication to having an MRI scan.

Absolute contra-indications to having an MRI scan include any shrapnel in the brain or eye in particular and certain cardiac valves and pacemakers

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Score (NRS) pain score: change in pain score over a follow-up period of 12 months: change in pain ratings as compared to pre-treatment ratings. | At 3 points during the 12 month follow-up: 1, 6 and 12 months after the last treatment
  This is the pain score the patient estimates he or she suffers from between 0 and 10. This is the pain score the patient estimates he or she suffers from between 0 and 10. An independent investigator contacts patients during the follow-up period and questions them about pain and function
Oxford Shoulder Score (OSS): change in function during a follow-up of 12 months as compared to pre-treatment scores | At 3 points during the 12 month follow-up: 1, 6 and 12 months after the last treatment
  This is a questionnaire evaluating function that may or may not be affected specifically by the affected shoulder.
Tear size as measured on MRI scanning | 6 after the last treatment
  Measurement of tear size on the MRI scan. The MRI scans are read by a musculoskeletal radiologist who is blinded to the treatment arm
Range of motion: change in range of motion over a period of 12 months as compared to pre-treatment scores. | 6 and 12 months after the last treatment
  Examination of passive range of motion of the shoulder. This is done by an independent researcher who is blinded to the treatment arm

CONTACTS AND LOCATIONS:
Locations (1):
- Pain Unit, Hadassah Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No